CLINICAL TRIAL: NCT07176494
Title: Revision of Deep Brain Stimulator in Patients With Parkinson's Disease: A Comparison of Perioperative Characteristics of Regional and General Anesthesia
Brief Title: Revision of Deep Brain Stimulator in Patients With Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, İbrahim Topcu, Principal Investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AnkaraEtlik1
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Pain Management; Regional Anesthesia; Deep Brain Stimulation; Parkinsons Disease
Keywords: Pectoserratus block; Interpektoral block; Deep brain stimulation; Awake surgery
MeSH Terms: conditions — Agnosia; Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who underwent surgery under general anesthesia (Active Comparator): These patients will be operated on under general anesthesia. During the skin closure, patients received 50 mg of dexketoprofen. Additionally, a paracetamol dose of 1 g every 8 hours and a dexketoprofen dose of 50 mg twice daily were administered intravenously for multimodal analgesia.
  Interventions: Procedure: Patients who underwent surgery under general anesthesia
- Patients who underwent surgery under regional anesthesia (Active Comparator): These patients will undergo surgery under regional anesthesia. Interpectoral and pectoserratus plane blocks will be applied to these patients. In the block group, bupivacaine and lidocaine are injected using an ultrasound-guided in-plane technique, between the 3rd and 4th ribs, into the interpectoral plane, and into the pectoserratus plane.
  25 cc (15 cc 0.5% bupivacaine + 5 cc 2% lidocaine + 5 cc isotonic) local anesthetic solution is prepared. 10 cc of the medication is administered into the interpectoral plane, and 15 cc into the pectoserratus plane.
  During the skin closure, patients received 50 mg of dexketoprofen. Additionally, a paracetamol dose of 1 g every 8 hours and a dexketoprofen dose of 50 mg twice daily were administered intravenously for multimodal analgesia.
  Interventions: Procedure: Patients who underwent surgery under regional anesthesia

INTERVENTIONS:
Procedure: Patients who underwent surgery under general anesthesia — Patients undergoing surgery under general anesthesia will undergo general anesthesia induction. During the skin closure, patients received 50 mg of dexketoprofen. Additionally, a paracetamol dose of 1 g every 8 hours and a dexketoprofen dose of 50 mg twice daily were administered intravenously for multimodal analgesia.
  Arms: Patients who underwent surgery under general anesthesia
Procedure: Patients who underwent surgery under regional anesthesia — 25 cc (15 cc 0.5% bupivacaine + 5 cc 2% lidocaine + 5 cc isotonic) local anesthetic solution is prepared. 10 cc of the medication is administered into the interpectoral plane, and 15 cc into the pectoserratus plane.
  During the skin closure, patients received 50 mg of dexketoprofen. Additionally, a paracetamol dose of 1 g every 8 hours and a dexketoprofen dose of 50 mg twice daily were administered intravenously for multimodal analgesia.
  Arms: Patients who underwent surgery under regional anesthesia

SUMMARY:
Parkinson's disease is a chronic and progressive neurodegenerative disease that affects the central nervous system, particularly impairing movement control. It is associated with the loss of dopamine-producing cells in the brain and typically occurs in middle age and beyond. Deep brain stimulation (DBS) is considered when symptoms of Parkinson's disease, such as tremors, slowed movements, and muscle rigidity, are not adequately controlled with medications. Selected patients with severe symptoms that do not respond to medical treatment are generally considered for this treatment.

Battery revision surgeries can be performed under general anesthesia or regional anesthesia. Patients undergoing general anesthesia should be cautious about the potential complications of general anesthesia, while those undergoing regional anesthesia should be cautious about the local anesthetic systemic toxicity. Because each method has its own advantages, the choice of anesthesia may vary.

This study aimed to compare postoperative analgesic efficacy and patient satisfaction in patients who underwent surgery under general anesthesia or sedation-assisted battery replacement under regional anesthesia. Both anesthesia methods are routinely used in Parkinson's disease patients undergoing battery replacement.

ELIGIBILITY:
Inclusion Criteria:

* Those aged 40-85
* Those with an ASA score of I-II-III
* Those with a body mass index (BMI) between 18-30

Exclusion Criteria:

* Those under 40 and over 85
* Those with an ASA score of IV or higher
* Those with a BMI of under 18 and over 30

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2026-07-05 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Pain score | up to 24 hours
  Pain will be assessed using a visual analog scale from 0 mm (no pain) to 100 mm (worst pain) at rest and when coughing. Pain assessment will be made at 0, 1, 6, 12, 18, and 24 hours after surgery.

SECONDARY OUTCOMES:
Patient Satisfaction | postoperative 24th hour
  Patient satisfaction will be evaluated using a Likert scale.Evaluation will be made using a 5-point Likert scale (1= I am not satisfied at all - 5= I am very satisfied).
Need for additional analgesics | postoperative 24th hour
  Additional analgesic need will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle\Ankara, Turkey (Türkiye)